CLINICAL TRIAL: NCT03268707
Title: Influence of an Innovative Telemetric Smartphone Application on Re-hospitalization And Quality of Life After Cryoballoon Pulmonary vEin Isolation in Patients With Paroxysmal Atrial Fibrillation
Brief Title: Influence of an Innovative Telemetric Smartphone Application on Re-hospitalization
Acronym: TRACE-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: PV5361
Record Dates: First submitted 2017-08-02; First posted 2017-08-31 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Paroxysmal Atrial Fibrillation; Pulmonary Vein Isolation; Telemetry Monitoring; Cryoballoon ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional follow up (Other): Conventional follow up at physician practice
  Interventions: Other: Conventional follow up
- Telemetric smartphone application (Experimental): Structured follow up with a telemetric smartphone application
  Interventions: Device: Telemetric smartphone application

INTERVENTIONS:
Device: Telemetric smartphone application — Structured follow up with a telemetric smartphone application
  Arms: Telemetric smartphone application
Other: Conventional follow up — Conventional follow up at physician practice
  Arms: Conventional follow up

SUMMARY:
A randomized, open, mono-centric pilot study to investigate the influence of an innovative telemetric smartphone application on re-hospitalization and quality of life after cryoballoon pulmonary vein isolation in patients with paroxysmal atrial fibrillation.

DETAILED DESCRIPTION:
The telemetric smartphone application includes a digitized medical record, a mobile ECG device and a 24-hour on call service by a cardiologist. The hypothesis is that the use of a telemetric smartphone application can reduce re-hospitalization in patients after cryoballoon pulmonary vein isolation. Secondary endpoints are quality of life measurements, health care cost calculations and recurrences of atrial fibrillation after ablation. All patients will undergo ablation and will be randomized into two groups: 1) conventional follow up with outpatient visits 6 and 12 months after ablation compared to 2) a structured follow up with the smartphone application, a mobile ECG device (patients will be able to send in as many ECGs as wanted), up to three phone calls with a cardiologist (24-hour on call service) as well as outpatient visits 6 and 12 months after cryo-ablation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Written informed consent
* symptomatic paroxysmal atrial fibrillation (at least two episodes within 3 months prior to ablation)
* cryoballoon pulmonary vein isolation
* possession of a compatible smartphone

Exclusion Criteria:

* Age < 18 years
* persistent or permanent atrial fibrillation (AF)
* prior catheter or surgical ablation of AF
* pregnant females
* contraindication for oral anticoagulation
* manifest hyper-/hypothyroidism
* no intention to cooperate
* alcoholism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-07-15 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Rehospitalization Recurrence of AF | in 12 months follow up
  Rate of rehospitalization after cryoballoon pulmonary vein isolation in patients with paroxysmal atrial fibrillation, Recurrence of sustained atrial fibrillation (>30 seconds) after atrial fibrillation ablation

CONTACTS AND LOCATIONS:
Overall Officials: Christian Meyer, MD, Principal Investigator — Universitaeres Herzzentrum Hamburg GmbH
Locations (2):
- Germany (2):
  - Asklepios St Georg, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg